CLINICAL TRIAL: NCT05481307
Title: An Open-label Phase 1 Study to Evaluate PK/PD Drug-drug Interactions and Safety/Tolerability Between RLD2202 and RLD2203 in Healthy Adult Subjects
Brief Title: A Study to Evaluate Pharmacokinetic/Pharmacodynamic Drug-drug Interaction and Safety/Tolerability Between RLD2202 and RLD2203
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HM-SARA-101
Record Dates: First submitted 2022-07-29; First posted 2022-08-01 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fixed Sequence (Experimental): Period 1: RLD2202, Period 2 : RLD2203 -> RLD2202+RLD2203
  Interventions: Drug: RLD2202; Drug: RLD2203

INTERVENTIONS:
Drug: RLD2202 — Take it once a day per period
Drug: RLD2203 — Take it once a day per period

SUMMARY:
The purpose of this study is to evaluate pharmacokinetic/pharmacodynamic drug-drug interactions and safety/tolerability between RLD2202 and RLD2203 in healthy adult subjects

ELIGIBILITY:
* Inclusion Criteria:

  1. Healthy adults in the age between 19 and 50 years old
  2. Body mass index (BMI) in the range of 18 to 27 kg/m2 and weight 50kg to 90kg.
  3. After fully hearing and understanding the details of this clinical trial, Subjects who have willingness to sign of informed consent before the screening.
  4. Subject who are eligible from physical examination, clinical laboratory test by investigators judgment.
* Exclusion Criteria:

  1. Presence of medical history or a concurrent disease that may interfere with treatment and safety assessment or completion of this clinical study, including clinically significant disorders in digestive system, neuropsychiatric system, endocrine system, liver, cardiovascular system
  2. Subjects who judged ineligible by the investigator

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2022-08-02 (Actual); Primary Completion 2022-10-25 (Actual); Study Completion 2022-10-25 (Actual)

PRIMARY OUTCOMES:
Cmax,ss of RLD2202 | 0~24 hours
  Pharmacokinetic evaluation
AUCtau,ss of RLD2202 | 0~24 hours
  Pharmacokinetic evaluation
Cmax,ss of RLD2203 | 0~24 hours
  Pharmacokinetic evaluation
AUCtau,ss of RLD2203 | 0~24 hours
  Pharmacokinetic evaluation
Inhibition of Platelet Aggregation(%) | 0~6 days
  Pharmacodynamic evaluation
Inhibition of Thromboxane B2(%) | 0~6 days
  Pharmacodynamic evaluation

SECONDARY OUTCOMES:
Tmax,ss of RLD2202 and RLD2203 | 0~24 hours
  Pharmacokinetic evaluation
t1/2,ss of RLD2202 and RLD2203 | 0~24 hours
  Pharmacokinetic evaluation
Cmin,ss of RLD2202 and RLD2203 | 0~24 hours
  Pharmacokinetic evaluation
Cavg,ss of RLD2202 and RLD2203 | 0~24 hours
  Pharmacokinetic evaluation
CLss/F of RLD2202 and RLD2203 | 0~24 hours
  Pharmacokinetic evaluation
Vdss/F of RLD2202 and RLD2203 | 0~24 hours
  Pharmacokinetic evaluation
PTF of RLD2202 and RLD2203 | 0~24 hours
  Pharmacokinetic evaluation

CONTACTS AND LOCATIONS:
Overall Officials: SeungHwan Lee, M.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea